CLINICAL TRIAL: NCT02763579
Title: A Phase I/III, Randomized, Double-Blind, Placebo-Controlled Study of Carboplatin Plus Etoposide With or Without Atezolizumab (Anti-PD-L1 Antibody) in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of Carboplatin Plus Etoposide With or Without Atezolizumab in Participants With Untreated Extensive-Stage (ES) Small Cell Lung Cancer (SCLC)
Acronym: IMpower133
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO30081; 2015-004861-97 (EudraCT Number)
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Atezolizumab + Carboplatin + Etoposide (Experimental): Participants received intravenous infusions of atezolizumab 1200 milligrams (mg) in combination with carboplatin to achieve an initial target area under the concentration-time curve (AUC) of 5 milligrams per milliliter per minute (mg/mL/min) followed by etoposide 100 milligrams per square meter (mg/m^2) on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) atezolizumab 1200 mg on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Carboplatin; Drug: Etoposide
- Placebo + Carboplatin + Etoposide (Active Comparator): Participants received intravenous infusions of placebo in combination with carboplatin to achieve an initial target AUC of 5 mg/mL/min followed by etoposide 100 mg/m^2 on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) placebo on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Placebo

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab intravenous infusion was administered at a dose of 1200 mg on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4) and maintenance phase (Cycle 5 onward).
  Other Names: MPDL3280A, RO5541267, Tecentriq
  Arms: Atezolizumab + Carboplatin + Etoposide
Drug: Carboplatin — Carboplatin intravenous infusion to achieve an initial target AUC of 5 mg/mL/min was administered on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4).
Drug: Etoposide — Etoposide intravenous infusion was administered at a dose of 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle during the induction phase (Cycles 1-4).
Drug: Placebo — Placebo intravenous infusion was administered on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4) and maintenance phase (Cycle 5 onward).
  Arms: Placebo + Carboplatin + Etoposide

SUMMARY:
This randomized, Phase I/III, multicenter, double-blinded, placebo-controlled study was designed to evaluate the safety and efficacy of atezolizumab (anti-programmed death-ligand 1 [PD-L1] antibody) in combination with carboplatin plus (+) etoposide compared with treatment with placebo + carboplatin + etoposide in chemotherapy-naive participants with ES-SCLC. Participants will be randomized in a 1:1 ratio to receive either atezolizumab + carboplatin + etoposide or placebo + carboplatin + etoposide on 21-day cycles for four cycles in the induction phase followed by maintenance with atezolizumab or placebo until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Treatment can be continued until persistent radiographic PD or symptomatic deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system)
* No prior systemic treatment for ES-SCLC
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function
* Treatment-free for at least 6 months since last chemo/radiotherapy, among those treated (with curative intent) with prior chemo/radiotherapy for limited-stage SCLC

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation
* Malignancies other than SCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Pregnant or lactating women
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Positive test result for human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C
* Severe infections at the time of randomization
* Significant cardiovascular disease
* Prior treatment with cluster of differentiation (CD) 137 agonists or immune checkpoint blockade therapies, anti-programmed death-1 (PD-1), and anti-PD-L1 therapeutic antibody
* History of severe (or known) hypersensitivity to chimeric or humanized antibodies or fusion proteins or any component of atezolizumab formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (114):
- United States (22):
  - Florida Cancer Specialists - Fort Myers (Broadway), Fort Myers, Florida
  - Florida Hospital, Orlando, Florida
  - Florida Cancer Specialists., St. Petersburg, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Cancer Treatment Centers of America - Midwestern Regional Medical Center, Zion, Illinois
  - Louisville Oncology, Louisville, Kentucky
  - New England Cancer Specialists, Scarborough, Maine
  - Weinberg CA Inst Franklin Sq, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - The Valley Hospital, Paramus, New Jersey
  - Broome Oncology - Binghamton, Binghamton, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology PLLC - Nashville (20th Ave), Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Prince Charles Hospital; Oncology Dept., Chermside, Queensland
  - Royal Melbourne Hospital; Hematology and Medical Oncology, Parkville, Victoria
- Austria (4):
  - Kepler Universitätskliniken GmbH - Med Campus III; Abt. für Lungenkrankheiten, Linz
  - Salzburger Landeskliniken; Universitätsklinik für Pneumologie/ Lungenheilkunde, Salzburg
  - Klinik Penzing; Abteilung für Atemwegs- und Lungenkrankheiten, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf; Abteilung Pulmologie, Vienna
- Brazil (4):
  - Santa Casa de Misericordia de Salvador, Salvador, Estado de Bahia
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Chile (2):
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - OrlandiOncología, Santiago
- China (9):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Na Bulovce, Prague
  - Thomayerova nemocnice, Praha 4 - Krc
- France (4):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Francois Baclesse; Oncologie, Caen
  - Hopital Calmette; Pneumologie Oncologie Ouest, Lille
  - Hôpital Nord - AP-HM Marseille#, Marseille
- Germany (5):
  - Asklepios-Fachklinik Muenchen-Gauting; Klinik Für Pneumologie, Gauting
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin II, Halle
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Fachklinik für Lungenerkrankungen, Immenhausen
- Greece (3):
  - Sotiria Chest Hospital of Athens, Athens
  - Agioi Anargyroi; 3Rd Dept. of Medical Oncology, Athens
  - University Hospital of Patras Medical Oncology, Pátrai
- Hungary (4):
  - Semmelweis Egyetem, AOK, Pulmonologiai Klinika, Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Tudogyogyaszati Klinika, Debrecen
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (6):
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - A.O. Universitaria Di Parma, Parma, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Irccs Istituto Europeo di Oncologia (IEO); Divisione di Oncologia, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Pisana - Ospedale Cisanello; Dipartimento Cardio Toraco Vascolare, Pisa, Tuscany
- Japan (13):
  - Kyushu University Hospital; Respiratory, Fukuoka
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Kanagawa Cancer Center;Thoracic Oncology, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine,?Pulmonary Medicine, Kyoto
  - Sendai Kousei Hospital; Pulmonary Medicine, Miyagi
  - Kurashiki Central Hospital; Respiratory Medicine, Okayama
  - Kindai University Hospital; Medical Oncology, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center; Internal Medicine, Osaka
  - Saitama Cancer Center; Thoracic Oncology, Satima
  - Shizuoka Cancer Center; Thoracic Oncology, Shizuoka
  - Tokyo Metropolitan Komagome Hospital; Thoracic Oncology and Respiratory Medicine, Tokyo
  - The Cancer Institute Hospital of JFCR, Respiratory Medicine, Tokyo
  - Wakayama Medical University Hospital; Respiratory Medicine and Medical Oncology, Wakayama
- Health Pharma Professional Research, Mexico City, Mexico CITY (federal District), Mexico
- Poland (6):
  - Medical University of Gdansk, Gdansk
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc; Oddzial V Chemioterapii Nowotworow Pluc, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
  - Centrum Onkologii - Inst.Im. Marii Sklodowskiej-Curie; Oncology, Warsaw
- Russia (6):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - N.N.Burdenko Main Military Clinical Hospital; Oncology Dept, Moscow, Moscow Oblast
  - Russian Oncology Research Center n.a. N.N. Blokhin, Moscow, Moscow Oblast
  - Scientific Research Oncology Institute named after N.N. Petrov; Oncology, Saint Petersburg, Sankt-Peterburg
  - City Clinical Onc., Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital No. 1, Novosibirsk
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Nis; Clinic for pulmonary diseases, Niš
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hosp Clinico Univ Lozano Blesa; División De Oncología Médica, Zaragoza
- Taiwan (3):
  - National Taiwan Uni Hospital; Internal Medicine, Taipei
  - Taipei Veterans General Hospital; Chest Dept , Section of Thoracic Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Chest Dept, Taoyuan District
- United Kingdom (4):
  - Royal Devon & Exeter Hospital; Oncology Centre, Exeter
  - Barts and the London NHS Trust., London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester

REFERENCES:
- [Derived] Bernabe R, Liu SV, Sanchez-Gastaldo A, Alonso Garcia M. Long-Term Survival and Stable Disease in a Patient with Extensive-Stage Small-Cell Lung Cancer after Treatment with Carboplatin, Etoposide and Atezolizumab. Oncol Ther. 2024 Mar;12(1):175-182. doi: 10.1007/s40487-023-00257-0. Epub 2024 Jan 27. PMID 38280181
- [Derived] Liu SV, Mok TSK, Nabet BY, Mansfield AS, De Boer R, Losonczy G, Sugawara S, Dziadziuszko R, Krzakowski M, Smolin A, Hochmair MJ, Garassino MC, Gay CM, Heymach JV, Byers LA, Lam S, Cardona A, Morris S, Adler L, Shames DS, Reck M. Clinical and molecular characterization of long-term survivors with extensive-stage small cell lung cancer treated with first-line atezolizumab plus carboplatin and etoposide. Lung Cancer. 2023 Dec;186:107418. doi: 10.1016/j.lungcan.2023.107418. Epub 2023 Oct 31. PMID 37931445
- [Derived] Liu SV, Reck M, Mansfield AS, Mok T, Scherpereel A, Reinmuth N, Garassino MC, De Castro Carpeno J, Califano R, Nishio M, Orlandi F, Alatorre-Alexander J, Leal T, Cheng Y, Lee JS, Lam S, McCleland M, Deng Y, Phan S, Horn L. Updated Overall Survival and PD-L1 Subgroup Analysis of Patients With Extensive-Stage Small-Cell Lung Cancer Treated With Atezolizumab, Carboplatin, and Etoposide (IMpower133). J Clin Oncol. 2021 Feb 20;39(6):619-630. doi: 10.1200/JCO.20.01055. Epub 2021 Jan 13. PMID 33439693
- [Derived] Mansfield AS, Kazarnowicz A, Karaseva N, Sanchez A, De Boer R, Andric Z, Reck M, Atagi S, Lee JS, Garassino M, Liu SV, Horn L, Wen X, Quach C, Yu W, Kabbinavar F, Lam S, Morris S, Califano R. Safety and patient-reported outcomes of atezolizumab, carboplatin, and etoposide in extensive-stage small-cell lung cancer (IMpower133): a randomized phase I/III trial. Ann Oncol. 2020 Feb;31(2):310-317. doi: 10.1016/j.annonc.2019.10.021. Epub 2019 Dec 9. PMID 31959349
- [Derived] Nishio M, Sugawara S, Atagi S, Akamatsu H, Sakai H, Okamoto I, Takayama K, Hayashi H, Nakagawa Y, Kawakami T. Subgroup Analysis of Japanese Patients in a Phase III Study of Atezolizumab in Extensive-stage Small-cell Lung Cancer (IMpower133). Clin Lung Cancer. 2019 Nov;20(6):469-476.e1. doi: 10.1016/j.cllc.2019.07.005. Epub 2019 Jul 31. PMID 31466854
- [Derived] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 114 centers in 21 countries: United States of America, Poland, Japan, Russia, Spain, Austria, Hungary, Czech Republic, South Korea, Italy, Serbia, Australia, Greece, United Kingdom, Germany, Taiwan, France, Chile, Brazil, Mexico, and China.
Pre-assignment Details: The total study population included 503 participants. The Global population included 403 participants. An additional 100 participants enrolled during the China Extension. The total China population included 10 Chinese participants from the Global population plus 100 participants from the China extension. 10 participants were part of the Global as well as China populations. Separate analyses were performed for the Global population and the China population in the study.
Groups:
- Placebo + Carboplatin + Etoposide - Global: Participants in the Global population received intravenous infusions of placebo in combination with carboplatin to achieve an initial target AUC of 5 mg/mL/min followed by etoposide 100 mg/m^2 on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) placebo on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
- Atezolizumab + Carboplatin + Etoposide - Global: Participants in the Global population received intravenous infusions of atezolizumab 1200 milligrams (mg) in combination with carboplatin to achieve an initial target area under the concentration-time curve (AUC) of 5 milligrams per milliliter per minute (mg/mL/min) followed by etoposide 100 milligrams per square meter (mg/m^2) on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) atezolizumab 1200 mg on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
- Placebo + Carboplatin + Etoposide - China: Participants in the China population received intravenous infusions of placebo in combination with carboplatin to achieve an initial target AUC of 5 mg/mL/min followed by etoposide 100 mg/m^2 on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) placebo on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
- Atezolizumab + Carboplatin + Etoposide - China: Participants in the China population received intravenous infusions of atezolizumab 1200 milligrams (mg) in combination with carboplatin to achieve an initial target area under the concentration-time curve (AUC) of 5 milligrams per milliliter per minute (mg/mL/min) followed by etoposide 100 milligrams per square meter (mg/m^2) on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) atezolizumab 1200 mg on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
Period: Global Period
Arm/Group | Placebo + Carboplatin + Etoposide - Global | Atezolizumab + Carboplatin + Etoposide - Global | Placebo + Carboplatin + Etoposide - China | Atezolizumab + Carboplatin + Etoposide - China
Started | 202 | 201 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 202 | 201 | 0 | 0
Not completed — Death | 167 | 151 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Study Terminated By Sponsor | 21 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 18 | 0 | 0
Period: China Period
Arm/Group | Placebo + Carboplatin + Etoposide - Global | Atezolizumab + Carboplatin + Etoposide - Global | Placebo + Carboplatin + Etoposide - China | Atezolizumab + Carboplatin + Etoposide - China
Started | 0 | 0 | 53 (n=4 Chinese participants from the Global population are included in the China population.) | 57 (n=6 Chinese participants from the Global population are included in the China population.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 53 | 57
Not completed — Death | 0 | 0 | 46 | 48
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Study Terminated By Sponsor | 0 | 0 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included 503 participants (All) with 403 in the Global population. An additional 100 participants enrolled in the China Extension. The China population included 10 Chinese participants from the Global population plus 100 participants from the China Extension. Separate analyses were performed for the Global population and the China population in the study.
Groups:
- Placebo + Carboplatin + Etoposide - All: All participants in the Global or China population received intravenous infusions of placebo in combination with carboplatin to achieve an initial target AUC of 5 mg/mL/min followed by etoposide 100 mg/m^2 on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) placebo on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
- Atezolizumab + Carboplatin + Etoposide - All: All participants in the Global or China population received intravenous infusions of atezolizumab 1200 milligrams (mg) in combination with carboplatin to achieve an initial target area under the concentration-time curve (AUC) of 5 milligrams per milliliter per minute (mg/mL/min) followed by etoposide 100 milligrams per square meter (mg/m^2) on Day 1 of every 21-day cycle during the induction phase (Cycles 1-4). On Days 2 and 3 of every 21-day cycle during the induction phase (Cycles 1-4), etoposide 100 mg/m^2 was administered alone. Thereafter, participants received maintenance (Cycle 5 onward) atezolizumab 1200 mg on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
- Total: Total of all reporting groups
Arm/Group | Placebo + Carboplatin + Etoposide - All | Atezolizumab + Carboplatin + Etoposide - All | Total
Number analyzed (Participants) | 251 | 252 | 503
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The intent-to-treat (ITT) population included 503 participants (All) with 403 in the Global population. An additional 100 participants enrolled in the China Extension. The China population included 10 Chinese participants from the Global population plus 100 participants from the China Extension.
  years
    Global: number analyzed (Participants) | 202 | 201 | 403
    Global | 63.6 (9.0) | 63.8 (8.8) | 63.7 (8.9)
    China: number analyzed (Participants) | 53 | 57 | 110
    China | 60.7 (8.8) | 59.7 (9.0) | 60.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants] — As reported from Electronic Case Report Form (eCRF). Population: The Global population included 403 participants. The China population included 100 participants enrolled during the China Extension plus 10 Chinese participants from the Global population.
  Participants
    Global: number analyzed (Participants) | 202 | 201 | 403
    Global: Female | 70 | 72 | 142
    Global: Male | 132 | 129 | 261
    China: number analyzed (Participants) | 53 | 57 | 110
    China: Female | 12 | 11 | 23
    China: Male | 41 | 46 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The intent-to-treat (ITT) population included 503 participants (All) with 403 in the Global population. An additional 100 participants enrolled in the China Extension. The China population included 10 Chinese participants from the Global population plus 100 participants from the China Extension.
  Participants
    Global: number analyzed (Participants) | 202 | 201 | 403
    Global: Hispanic or Latino | 8 | 8 | 16
    Global: Not Hispanic or Latino | 185 | 187 | 372
    Global: Unknown or Not Reported | 9 | 6 | 15
    China: number analyzed (Participants) | 53 | 57 | 110
    China: Hispanic or Latino | 0 | 0 | 0
    China: Not Hispanic or Latino | 53 | 57 | 110
    China: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The intent-to-treat (ITT) population included 503 participants (All) with 403 in the Global population. An additional 100 participants enrolled in the China Extension. The China population included 10 Chinese participants from the Global population plus 100 participants from the China Extension.
  Participants
    Global: number analyzed (Participants) | 202 | 201 | 403
    Global: American Indian or Alaska Native | 1 | 0 | 1
    Global: Asian | 36 | 33 | 69
    Global: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Global: Black or African American | 2 | 1 | 3
    Global: White | 159 | 163 | 322
    Global: More than one race | 0 | 0 | 0
    Global: Unknown or Not Reported | 4 | 4 | 8
    China: number analyzed (Participants) | 53 | 57 | 110
    China: American Indian or Alaska Native | 0 | 0 | 0
    China: Asian | 53 | 57 | 110
    China: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    China: Black or African American | 0 | 0 | 0
    China: White | 0 | 0 | 0
    China: More than one race | 0 | 0 | 0
    China: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration of Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1 in the Global Population
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least 20% increase in the sum of the longest diameter of target lesions compared to baseline, or unequivocal progression in non-target lesion(s), or the appearance of new lesion(s).
Time Frame: Baseline until PD or death, whichever occurs first (up to approximately 23 months)
Population: The ITT population was defined as all randomized participants, regardless of whether the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 202 | 201
Months | 4.3 (4.2) [4.2 to 4.5] | 5.2 (4.4) [4.4 to 5.6]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.0170, Log Rank; Stratified Hazard Ratio = 0.77, 95% CI 2-sided [0.62 to 0.96]

2. Primary Outcome: Duration of Overall Survival (OS) in the Global Population
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: Baseline until death from any cause (up to approximately 23 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 202 | 201
Months | 10.3 (9.3) [9.3 to 11.3] | 12.3 (10.8) [10.8 to 15.9]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.0069, Log Rank; Stratified Hazard Ratio = 0.70, 95% CI 2-sided [0.54 to 0.91]

3. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) as Assessed by the Investigator Using RECIST v1.1 in the Global Population
Description: Objective response (OR) is defined as complete response (CR) or partial response (PR) as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline until partial response (PR) or complete response (CR), whichever occurs first (up to approximately 23 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 202 | 201
Percentage of participants | 76.7 [70.29 to 82.38] | 74.1 [67.50 to 80.03]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.55 to 1.37]

4. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator Using RECIST v1.1 in the Global Population
Description: DOR is defined as the time interval from first occurrence of a documented objective response to the time of disease progression as determined by the investigator using RECIST v1.1 or death from any cause, whichever comes first.
Time Frame: First occurrence of PR or CR until PD or death, whichever occurs first (up to approximately 23 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 155 | 149
Months | 3.1 [2.9 to 3.9] | 4.1 [3.5 to 4.2]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.0063, Log Rank; Hazard Ratio (HR) = 0.715, 95% CI 2-sided [0.562 to 0.911]

5. Secondary Outcome: PFS Rate at 6 Months and at 1 Year in Global Population
Description: PFS rates at 6 months and at 1 year is defined as the proportion of participants who are alive without disease progression 6 months and 1 year after randomization, respectively.
Time Frame: 6 months, 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 202 | 201
Percentage of participants
  6 Months | 22.39 [16.56 to 28.22] | 30.86 [24.26 to 37.45]
  1 Year | 5.35 [2.14 to 8.56] | 12.62 [7.85 to 17.40]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; PFS Rate at 6 months; Test type: Superiority; p = 0.0593, Z-test; Difference in Event Free Rate = 8.47, 95% CI 2-sided [-0.33 to 17.27]
Statistical Analysis 2: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; PFS Rate at 1 year; Test type: Superiority; p = 0.0133, Z-test; Difference in Event Free Rate = 7.27, 95% CI 2-sided [1.52 to 13.02]

6. Secondary Outcome: OS Rate at 1 Year and 2 Years in the Global Population
Description: OS rates at 1 and 2 years is defined as the proportion of participants who are alive 1 year and 2 years after randomization, respectively.
Time Frame: 1 year, 2 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 202 | 201
Percentage of participants
  1 Year | 38.23 | 51.69
  2 Years | NA — Insufficient number of participants with events. | NA — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; OS Rate at 1 year; Test type: Superiority; p = 0.0095, Z-test; Difference in Event Free Rate = 13.46, 95% CI 2-sided [3.29 to 23.64]

7. Secondary Outcome: Time to Deterioration (TTD) Per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 (C30) and Supplemental Lung Cancer Module (QLQ-LC13) in the Global Population
Description: TTD according to the EORTC QLQ-C30 and EORTC QLQ-LC13 measures were evaluated in each of the following linearly transformed symptom scores: cough, dyspnea (single item), dyspnea (multi-item subscale), chest pain, or arm/shoulder pain. The linear transformation gives each individual symptom subscale a possible score of 0 to 100. For the symptom to be considered "deteriorated," a score increase of ≥10 points above baseline must be held for at least two consecutive assessments or an initial score increase of ≥10 points is followed by death within 3 weeks from the last assessment. A ≥ 10-point change in the symptoms subscale score is perceived by participants as clinically significant.
Time Frame: Baseline until deterioration per symptom subscale (up to approximately 23 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 202 | 201
Month
  Cough | NA [16.6 to NA] — Insufficient number of participants with events. | 20.3 [NA to NA] — Insufficient number of participants with events.
  Pain in Chest | NA [10.9 to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.
  Pain in Arm or Shoulder | NA [8.8 to NA] — Insufficient number of participants with events. | NA [9.2 to NA] — Insufficient number of participants with events.
  Dyspnea | 5.6 [3.6 to 8.8] | NA [5.5 to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Cough; Test type: Superiority — Stratified analysis. Stratification factors: Sex (male vs female) and ECOG (0 vs 1); p = 0.3604, Log Rank; Hazard Ratio (HR) = 1.221, 95% CI 2-sided [0.795 to 1.874]
Statistical Analysis 2: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Pain in Chest; Test type: Superiority — Stratified analysis. Stratification factors: Sex (male vs female) and ECOG (0 vs 1); p = 0.7712, Log Rank; Hazard Ratio (HR) = 1.058, 95% CI 2-sided [0.722 to 1.553]
Statistical Analysis 3: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Pain in Arm or Shoulder; Test type: Superiority — Stratified analysis. Stratification factors: Sex (male vs female) and ECOG (0 vs 1); p = 0.6922, Log Rank; Hazard Ratio (HR) = 1.077, 95% CI 2-sided [0.747 to 1.552]
Statistical Analysis 4: Comparison: Placebo + Carboplatin + Etoposide vs Atezolizumab + Carboplatin + Etoposide; Dyspnea; Test type: Superiority — Stratified analysis. Stratification factors: Sex (male vs female) and ECOG (0 vs 1); p = 0.0650, Log Rank; Hazard Ratio (HR) = 0.748, 95% CI 2-sided [0.549 to 1.019]

8. Secondary Outcome: Percentage of Participants With at Least One Adverse Event in the Global Population
Description: The percentage of participants with at least one adverse event in the global population.
Time Frame: Baseline until up to 90 days after end of treatment (up to approximately 49 months)
Population: The safety population included all treated participants, defined as participants who received any amount of any component of study treatment. For the safety analyses, patrticipants who received any amount of atezolizumab were analyzed as part of the Atezo + CE arm, even if atezolizumab was given in error.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 196 | 198
Percentage of participants | 96.4 | 100.0

9. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) to Atezolizumab in the Global Population
Description: The baseline prevalence and post-baseline incidence of ADAs against atezolizumab.
Time Frame: Predose (0 hours [H]) on Day (D) 1 of Cycles (C) 1, 2, 3, 4, 8, 16, and every 8 cycles (Q8C) thereafter (cycle = 21 days) until treatment discontinuation (up to 23 months) and 120 days after last dose (up to approximately 23 months overall)
Population: ADA analyses were based on ADA observations from participants who had received atezolizumab treatment and were evaluated for immunogenicity.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 198
Percentage of participants
  Baseline evaluable participants: number analyzed (Participants) | 196
  Baseline evaluable participants | 2.0
  Post-baseline evaluable participants: number analyzed (Participants) | 188
  Post-baseline evaluable participants | 18.6

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Atezolizumab in the Global Population
Description: Atezolizumab maximum observed plasma concentration (Cmax; 30 minutes following the end of the atezolizumab infusion) for each respective day.
Time Frame: Post-dose Day 1 of Cycle 1 (cycle length = 21 days)
Population: PK analyses were based on PK observations from all participants who had received atezolizumab, carboplatin, or etoposide treatment and who provided at least one evaluable atezolizumab PK sample.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 185
μg/mL | 389 (135)

11. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Atezolizumab in the Global Population
Description: Atezolizumab pre-dose plasma concentration (Cmin) for each respective day.
Time Frame: Predose on Day 1 of Cycles 1, 3, 4, 8, 16 and 24 (cycle length = 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 194
μg/mL
  Cycle 1 Day 1 | NA (NA) — Below the level of detection.
  Cycle 3 Day1: number analyzed (Participants) | 174
  Cycle 3 Day1 | 80.6 (32.1)
  Cycle 4 Day 1: number analyzed (Participants) | 156
  Cycle 4 Day 1 | 138 (56.4)
  Cycle 8 Day 1: number analyzed (Participants) | 88
  Cycle 8 Day 1 | 186 (73.5)
  Cycle 16 Day 1: number analyzed (Participants) | 22
  Cycle 16 Day 1 | 196 (63.1)
  Cycle 24 Day 1: number analyzed (Participants) | 4
  Cycle 24 Day 1 | 221 (43.4)

12. Secondary Outcome: Plasma Concentration of Carboplatin in the Global Population
Description: Plasma concentration of carboplatin in the Global population.
Time Frame: Predose, before end of infusion, and after end of carboplatin infusion on Day 1 of Cycle 1 and Cycle 3 (cycle = 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 13 | 13
ng/mL
  Pre-Dose on Day 1 of Cycle 1: number analyzed (Participants) | 12 | 11
  Pre-Dose on Day 1 of Cycle 1 | NA (NA) — Below level of detection. | NA (NA) — Below level of detection.
  Before End of Infusion on Day 1 of Cycle 1: number analyzed (Participants) | 12 | 11
  Before End of Infusion on Day 1 of Cycle 1 | 13300 (4880) | 11200 (5060)
  Post Infusion on Day 1 of Cycle 1: number analyzed (Participants) | 11 | 12
  Post Infusion on Day 1 of Cycle 1 | 7200 (1880) | 6860 (1670)
  Pre-Dose on Day 1 of Cycle 3: number analyzed (Participants) | 12 | 13
  Pre-Dose on Day 1 of Cycle 3 | 144 (58.3) | 126 (48.1)
  Before End of Infusion on Day 1 of Cycle 3 | 13900 (3590) | 11300 (5090)
  Post Infusion on Day 1 of Cycle 3 | 7180 (1630) | 6540 (2200)

13. Secondary Outcome: Plasma Concentration of Etoposide in the Global Population
Description: Plasma concentration of etoposide in the Global Population.
Time Frame: Predose, before end of infusion, 1 and 4 hours after end of carboplatin infusion on Day 1 of Cycle 1 and Cycle 3 (cycle = 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo + Carboplatin + Etoposide | Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 13 | 13
ng/mL
  Pre-Dose on Day 1 of Cycle 1: number analyzed (Participants) | 12 | 13
  Pre-Dose on Day 1 of Cycle 1 | NA (NA) — Below level of detection. | NA (NA) — Below level of detection.
  Before End of Infusion on Day 1 of Cycle 1: number analyzed (Participants) | 10 | 10
  Before End of Infusion on Day 1 of Cycle 1 | 17000 (3640) | 19400 (2860)
  1 Hour Post Infusion on Day 1 of Cycle 1: number analyzed (Participants) | 8 | 12
  1 Hour Post Infusion on Day 1 of Cycle 1 | 11100 (2010) | 12600 (1960)
  4 Hours Post Infusion on Day 1 of Cycle 1: number analyzed (Participants) | 9 | 9
  4 Hours Post Infusion on Day 1 of Cycle 1 | 7640 (2360) | 7300 (1230)
  Pre-Dose on Day 1 of Cycle 3 | NA (NA) — Below level of detection. | NA (NA) — Below level of detection.
  Before End of Infusion on Day 1 of Cycle 3: number analyzed (Participants) | 11 | 9
  Before End of Infusion on Day 1 of Cycle 3 | 16600 (2180) | 17700 (3600)
  1 Hour Post Infusion on Day 1 of Cycle 3: number analyzed (Participants) | 10 | 13
  1 Hour Post Infusion on Day 1 of Cycle 3 | 12400 (3740) | 12200 (2810)
  4 Hours Post Infusion on Day 1 of Cycle 3: number analyzed (Participants) | 10 | 11
  4 Hours Post Infusion on Day 1 of Cycle 3 | 6740 (1230) | 7960 (2090)

ADVERSE EVENTS:
Time Frame: From the first study drug administration to the data cutoff date: 7 July 2022 (up to 49 months).
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. Serious & other adverse events reported based on safety population, which included participants who received any amount of any component of study treatment.
Arm/Group | Placebo + Carboplatin + Etoposide - Global | Atezolizumab + Carboplatin + Etoposide - Global | Placebo + Carboplatin + Etoposide - China | Atezolizumab + Carboplatin + Etoposide - China
All-Cause Mortality (participants affected / at risk) | 11/196 | 5/198 | 1/52 | 3/57
Serious Adverse Events (participants affected / at risk) | 69/196 | 81/198 | 14/52 | 22/57
Other Adverse Events (participants affected / at risk) | 187/196 | 191/198 | 52/52 | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Carboplatin + Etoposide - Global (N=196) | Atezolizumab + Carboplatin + Etoposide - Global (N=198) | Placebo + Carboplatin + Etoposide - China (N=52) | Atezolizumab + Carboplatin + Etoposide - China (N=57)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 5 (5) | 2 (2) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 7 (7) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 10 (11) | 12 (15) | 4 (5) | 4 (7)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyopneumothorax (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Carboplatin + Etoposide - Global (N=196) | Atezolizumab + Carboplatin + Etoposide - Global (N=198) | Placebo + Carboplatin + Etoposide - China (N=52) | Atezolizumab + Carboplatin + Etoposide - China (N=57)
Anaemia (Blood and lymphatic system disorders) | 69 (84) | 86 (101) | 40 (50) | 46 (76)
Leukopenia (Blood and lymphatic system disorders) | 19 (32) | 24 (44) | 14 (22) | 9 (24)
Neutropenia (Blood and lymphatic system disorders) | 66 (105) | 71 (122) | 17 (41) | 11 (32)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (44) | 31 (46) | 16 (31) | 17 (27)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 2 (2) | 4 (4) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 5 (5) | 11 (11) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 20 (20) | 2 (2) | 8 (9)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 10 (10) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 58 (70) | 52 (65) | 8 (12) | 10 (19)
Diarrhoea (Gastrointestinal disorders) | 30 (46) | 34 (46) | 2 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 65 (95) | 77 (112) | 10 (15) | 21 (47)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 11 (11) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 34 (49) | 40 (52) | 7 (7) | 14 (20)
Asthenia (General disorders) | 20 (26) | 25 (29) | 4 (5) | 4 (4)
Chest discomfort (General disorders) | 5 (5) | 2 (2) | 2 (2) | 5 (5)
Chest pain (General disorders) | 14 (14) | 18 (22) | 4 (4) | 5 (5)
Fatigue (General disorders) | 51 (67) | 52 (66) | 0 (0) | 6 (8)
Oedema peripheral (General disorders) | 7 (8) | 13 (14) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 16 (18) | 20 (32) | 4 (7) | 13 (19)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (5) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 17 (20) | 15 (19) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (6) | 13 (18) | 5 (5) | 2 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (9) | 10 (13) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (6) | 6 (13) | 10 (15) | 13 (21)
Aspartate aminotransferase increased (Investigations) | 5 (7) | 8 (9) | 9 (16) | 11 (15)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 8 (8) | 3 (4) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 5 (6) | 2 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 8 (23)
Blood creatinine increased (Investigations) | 3 (3) | 7 (13) | 3 (3) | 4 (8)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 4 (5) | 6 (18)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (4) | 4 (4) | 2 (2)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 4 (6)
Neutrophil count decreased (Investigations) | 45 (80) | 37 (74) | 33 (85) | 41 (107)
Platelet count decreased (Investigations) | 30 (41) | 26 (38) | 14 (26) | 24 (40)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Weight decreased (Investigations) | 10 (11) | 21 (21) | 6 (6) | 10 (10)
Weight increased (Investigations) | 6 (7) | 3 (3) | 4 (4) | 1 (1)
White blood cell count decreased (Investigations) | 24 (43) | 18 (35) | 29 (73) | 34 (101)
Decreased appetite (Metabolism and nutrition disorders) | 41 (45) | 55 (64) | 12 (16) | 13 (22)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (7) | 9 (13) | 2 (3) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5) | 5 (5) | 9 (14)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 4 (7) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (18) | 9 (9) | 5 (10) | 5 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (10) | 13 (19) | 2 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (14) | 10 (10) | 11 (17) | 10 (12)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (29) | 25 (31) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (20) | 19 (19) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 13 (13) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 11 (14) | 20 (23) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 23 (26) | 25 (30) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 14 (14) | 16 (19) | 3 (9) | 4 (8)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 7 (10) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (33) | 22 (28) | 10 (12) | 14 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 21 (24) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 14 (20) | 5 (6) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 13 (17) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 10 (10) | 5 (5) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 69 (72) | 73 (75) | 18 (18) | 25 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 15 (17) | 1 (1) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 13 (15) | 15 (25) | 1 (1) | 6 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 11 (11) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (8) | 15 (20) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT02763579/Prot_SAP_000.pdf